CLINICAL TRIAL: NCT04263688
Title: Multicenter Observational Study for Correlation Between Tumor Mutation Burden and Immunotherapy Efficacy of Advanced Non-small Cell Lung Cancer With Malignant Pleural Effusion
Brief Title: Multicenter Observational Study of Advanced Non-small Cell Lung Cancer With Malignant Pleural Effusion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, Chief Physician, Guangzhou Institute of Respiratory Disease
Other Study IDs: LC-IMMA
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Multicenter Observational Study; Tumor Mutation Burden (TMB); immunotherapy; Pleural effusion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunotherapy effective: Immunotherapy was applied for 8 weeks to evaluate the efficacy，The efficacy of immunotherapy was evaluated by imaging, and was evaluated according to RECIST 1.1.
  Interventions: Other: Non-Intervention
- Immunotherapy Ineffective: Immunotherapy was applied for 8 weeks to evaluate the efficacy，The efficacy of immunotherapy was evaluated by imaging, and was evaluated according to RECIST 1.1.
  Interventions: Other: Non-Intervention

INTERVENTIONS:
Other: Non-Intervention — Non-Intervention

SUMMARY:
Multicenter observational study for correlation between tumor mutation burden and immunotherapy efficacy of advanced non-small cell lung cancer with malignant pleural effusion

DETAILED DESCRIPTION:
Method of Research:

1. ⅢB-Ⅳ NSCLC patients, tumor mutation burden (TMB) was tested by the 448 gene panel with pleural effusion and tissue sample, to observed mutation characteristics;Tissue and pleural effusion cell precipitation:TMB (Next generation sequencing, 448 gene panel;Average sequencing depth: above 5000×)
2. The date of blood routine examination(neutrophils to lymphocytes ratio (NLR)) and serological tumor maker of NSCLC were collected before treatment;the The results of Programmed death ligand 1 (PDL1) expression level were collected also;
3. Collected Imaging(CT)and pathological data before treatment;
4. Immunotherapy was applied for 8 weeks to evaluate the efficacy;
5. The tumor mutation burden of pleural effusion was tested again for the patients of hyper-progression after immunotherapy, the mutation characteristics and changes were observed, the molecular mutation change before and after treatment were evaluated, and the correlation with immunotherapy was analyzed.Hyper-progression (HPD) were defined as tumor growth rate excess of 50% compared to baseline CT scans prior to treatment initiation.The patient underwent imaging examination (chest CT or pet-ct) at 2 months (8 weeks) after 3 full doses of immunotherapy drugs.
6. The date of blood routine examination(neutrophils to lymphocytes ratio (NLR)) and serological tumor maker of NSCLC were collected after treatment;
7. Imaging, CT and pathological data of patients after treatment were collected

ELIGIBILITY:
Inclusion Criteria:

1. male or female,18 years ≤ age ≤80 years;
2. Pathologically confirmed stage ⅢB-Ⅳ NSCLC, which is not suitable for surgical resection;
3. No systematic anti-tumor treatment;
4. Pleural effusion ≥50ml,tissue samples can be obtained;
5. The driver gene was negative, and immunotherapy was proposed;
6. According to RECIST 1.1, at least one tumor lesion that can be measured or evaluated;
7. Signed and dated informed consent

Exclusion Criteria:

1. No pathological diagnosis or the diagnosis is not clear;
2. Severe pneumonia or tuberculosis;
3. Tumor tissues cannot be obtained;
4. Combine with other tumor type or other subtypes of lung cancer;
5. Poor compliance, unable to complete follow-up;
6. The investigator judges the situation that may affect the clinical search process and results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically proven diagnosis of ⅢB-Ⅳ NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) of NSCLC patients with malignant pleural effusion who were received immunotherapy | 2021
  The relationship between tumor mutation burden and objective response rate in NSCLC patients
Progression-free survival (PFS) of NSCLC patients with malignant pleural effusion who were received immunotherapy | 2021
  The relationship between tumor mutation burden and progression-free survival in NSCLC patients
Overall survival (OS) of NSCLC patients with malignant pleural effusion who were received immunotherapy | 2022
  The relationship between tumor mutation burden and overall survival in NSCLC patients

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gandara DR, Paul SM, Kowanetz M, Schleifman E, Zou W, Li Y, Rittmeyer A, Fehrenbacher L, Otto G, Malboeuf C, Lieber DS, Lipson D, Silterra J, Amler L, Riehl T, Cummings CA, Hegde PS, Sandler A, Ballinger M, Fabrizio D, Mok T, Shames DS. Blood-based tumor mutational burden as a predictor of clinical benefit in non-small-cell lung cancer patients treated with atezolizumab. Nat Med. 2018 Sep;24(9):1441-1448. doi: 10.1038/s41591-018-0134-3. Epub 2018 Aug 6. PMID 30082870
- [Background] Qin BD, Jiao XD, Zang YS. Tumor mutation burden to tumor burden ratio and prediction of clinical benefit of anti-PD-1/PD-L1 immunotherapy. Med Hypotheses. 2018 Jul;116:111-113. doi: 10.1016/j.mehy.2018.05.005. Epub 2018 May 16. PMID 29857892
- [Background] Samstein RM, Lee CH, Shoushtari AN, Hellmann MD, Shen R, Janjigian YY, Barron DA, Zehir A, Jordan EJ, Omuro A, Kaley TJ, Kendall SM, Motzer RJ, Hakimi AA, Voss MH, Russo P, Rosenberg J, Iyer G, Bochner BH, Bajorin DF, Al-Ahmadie HA, Chaft JE, Rudin CM, Riely GJ, Baxi S, Ho AL, Wong RJ, Pfister DG, Wolchok JD, Barker CA, Gutin PH, Brennan CW, Tabar V, Mellinghoff IK, DeAngelis LM, Ariyan CE, Lee N, Tap WD, Gounder MM, D'Angelo SP, Saltz L, Stadler ZK, Scher HI, Baselga J, Razavi P, Klebanoff CA, Yaeger R, Segal NH, Ku GY, DeMatteo RP, Ladanyi M, Rizvi NA, Berger MF, Riaz N, Solit DB, Chan TA, Morris LGT. Tumor mutational load predicts survival after immunotherapy across multiple cancer types. Nat Genet. 2019 Feb;51(2):202-206. doi: 10.1038/s41588-018-0312-8. Epub 2019 Jan 14. PMID 30643254
- [Background] Chalmers ZR, Connelly CF, Fabrizio D, Gay L, Ali SM, Ennis R, Schrock A, Campbell B, Shlien A, Chmielecki J, Huang F, He Y, Sun J, Tabori U, Kennedy M, Lieber DS, Roels S, White J, Otto GA, Ross JS, Garraway L, Miller VA, Stephens PJ, Frampton GM. Analysis of 100,000 human cancer genomes reveals the landscape of tumor mutational burden. Genome Med. 2017 Apr 19;9(1):34. doi: 10.1186/s13073-017-0424-2. PMID 28420421
- [Background] Wang Z, Duan J, Cai S, Han M, Dong H, Zhao J, Zhu B, Wang S, Zhuo M, Sun J, Wang Q, Bai H, Han J, Tian Y, Lu J, Xu T, Zhao X, Wang G, Cao X, Li F, Wang D, Chen Y, Bai Y, Zhao J, Zhao Z, Zhang Y, Xiong L, He J, Gao S, Wang J. Assessment of Blood Tumor Mutational Burden as a Potential Biomarker for Immunotherapy in Patients With Non-Small Cell Lung Cancer With Use of a Next-Generation Sequencing Cancer Gene Panel. JAMA Oncol. 2019 May 1;5(5):696-702. doi: 10.1001/jamaoncol.2018.7098. PMID 30816954
- [Background] Yarchoan M, Hopkins A, Jaffee EM. Tumor Mutational Burden and Response Rate to PD-1 Inhibition. N Engl J Med. 2017 Dec 21;377(25):2500-2501. doi: 10.1056/NEJMc1713444. No abstract available. PMID 29262275